CLINICAL TRIAL: NCT03570723
Title: Glove-loaded Foley's Catheter Tamponade to Reducing Blood Loss During Cesarean Delivery for Complete Placenta Previa: a Randomized Controlled Trial
Brief Title: Glove-loaded Foley's Catheter Tamponade for Cesarean Section for Placenta Previa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, lecturer, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: aswu/201/18
Record Dates: First submitted 2018-05-06; First posted 2018-06-27 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Placenta Previa; Post Partum Hemorrhage
MeSH Terms: conditions — Placenta Previa; Postpartum Hemorrhage

STUDY DESIGN:
Intervention Model Description: The study was single-blind randomized controlled trial carried out in a tertiary University Hospital between June 2018to June 2021. Investigators included patients scheduled for CS due to complete placenta previa. They were randomly allocated to the group (I) managed by stepwise uterine devascularization, group (II) managed by A glove-loaded Foley's catheter tamponade. The primary outcome was the amount of intraoperative estimated blood loss.
Who Masked: Participant
Masking Description: The participants were blinded to the procedure performed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stepwise uterine devascularization (Active Comparator): Uterine hemostatic sutures, through examination of the placental bed, may use some hemostasis at the placental bed,"overswing" was commenced using endo-uterine sutures. If there is still significant bleeding, bilateral uterine artery ligation, and internal iliac artery ligation when needed.BUAL started immediately through blunt dissection downwards and laterally of the peritoneum covering the uterine isthmus and cervix. The peritoneum is mobilized freely at the uterine angles to expose both uterine arteries and avoid inclusion of the ureters in the ligation. The uterine artery pulsations were palpated digitally at the level of the internal os.
  Interventions: Procedure: stepwise uterine devascularization
- A glove-loaded Foley's catheter (Experimental): A glove-loaded Foley's catheter tamponade, the internal os of the cervix was identified and a double-way 20 Fr Foley's catheter with a 30-50-ml balloon was inserted through the cervix to be handled by an assistant through the vagina and fixed to the patient's lower limb after inflation of the catheter balloon by 300 ml warm saline and pulling it against the lower uterine segment between the two transverse sutures. Only one glove-loaded Foley's catheter was used for tamponade.
  Interventions: Procedure: A glove-loaded Foley's catheter tamponade

INTERVENTIONS:
Procedure: A glove-loaded Foley's catheter tamponade — A glove-loaded Foley's catheter tamponade, the internal os of the cervix was identified and a double-way 20 Fr Foley's catheter with a 30-50-ml balloon was inserted through the cervix to be handled by an assistant through the vagina and fixed to the patient's lower limb after inflation of the catheter balloon by 300 ml warm saline and pulling it against the lower uterine segment between the two transverse sutures. Only one glove-loaded Foley's catheter was used for tamponade.
  Other Names: Foley's tamponade
  Arms: A glove-loaded Foley's catheter
Procedure: stepwise uterine devascularization — Uterine hemostatic sutures, through examination of the placental bed, may use some hemostasis at the placental bed,"overswing" was commenced using endo-uterine sutures. If there is still significant bleeding, bilateral uterine artery ligation, and internal iliac artery ligation when needed.BUAL started immediately through blunt dissection downwards and laterally of the peritoneum covering the uterine isthmus and cervix. The peritoneum is mobilized freely at the uterine angles to expose both uterine arteries and avoid inclusion of the ureters in the ligation. The uterine artery pulsations were palpated digitally at the level of the internal os.
  Arms: stepwise uterine devascularization

SUMMARY:
Objective: To investigate the effect of A glove-loaded Foley's catheter tamponade versus stepwise uterine devascularization on blood loss during cesarean section (CS) in patients with complete placenta previa.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) due to placenta previa is usually from the placental bed at the lower uterine segment and it occurs after the placenta separation.

Despite placenta previa can be diagnosed by obstetrician before delivery nowadays, still a leading etiology of maternal mortality and morbidity.

Placenta previa is an obstetric condition that is closely linked with massive obstetric hemorrhage. Is not only associated with increased chance of requiring massive transfusion (> 3 units of packed red blood cells) but also a is now the leading etiology of the cesarean hysterectomies. The incidence has progressively risen worldwide, mainly due to the increasing rates of cesarean section.

Uterine tamponade can be considered as a line of treatment before performing surgical procedures in PPH resulting from the placental site bleeding. It can save the life, avoid laparotomy and preserve fertility.

Nowadays, the use of intrauterine balloons has been developed and become effective for the control of placental site bleeding not responding to medical treatment.

The 2-way Foley's catheter has many advantages over the gauze packing; first, it allows drainage of blood, so no occult bleeding could be accumulated inside the uterus as in uterine gauze, second the removal of the Foley's catheter balloon is easy and not painful, third, the removal of 2-way Foley's catheter could be gradual as a test of its effectiveness before complete removal.

Bakri intrauterine balloon tamponade is used for the treatment of obstetric hemorrhage during cesarean delivery and many recent reports had described the successful use of balloon tamponade to manage hemorrhage due to placenta previa- with an overall success rate of 80%. However; its price is high so in our country, its availability and use are difficult.

So, the aims of this study to assess the effect of A glove-loaded Foley's catheter tamponade versus stepwise uterine devascularization on blood loss during cesarean section (CS) in patients with complete placenta previa.

The study will be single blinded randomized controlled trial carried out in a tertiary University Hospital between June 2018to June 2021. The included patients will be scheduled for CS due to complete placenta previa. They will be randomly allocated to the group (I) managed by stepwise uterine devascularization, group (II) managed by A glove-loaded Foley's catheter tamponade. The primary outcome will be the amount of intraoperative estimated blood loss.

ELIGIBILITY:
Inclusion Criteria:

* all pregnant women with a single-term fetus scheduled for elective CD for complete placenta previa

Exclusion Criteria:

* • Patients with the cardiac, hepatic, renal, or thromboembolic disease;

  * patients with the high possibility of morbid adherent placenta;
  * known coagulopathy, and
  * those presented with severe antepartum hemorrhage were excluded.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
intraoperative blood loss | during the operation
  blood loss during operation

SECONDARY OUTCOMES:
cesarean hysterectomy | intraoperative
  cesarean hysterectomy
need for blood transfusion | intraoperative and post operative 4 hours blood loss estimation
  need for blood transfusion
postoperative blood loss | 4 hours post operative
  blood loss post operative

CONTACTS AND LOCATIONS:
Locations (1):
- AswanUH, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kellie FJ, Wandabwa JN, Mousa HA, Weeks AD. Mechanical and surgical interventions for treating primary postpartum haemorrhage. Cochrane Database Syst Rev. 2020 Jul 1;7(7):CD013663. doi: 10.1002/14651858.CD013663. PMID 32609374